CLINICAL TRIAL: NCT00190502
Title: The Use of Polyclonal Anti-T-Lymphocyte Globulin to Prevent Progression of Autoimmune Beta-Cell Destruction in Recent Type 1 Diabetes
Brief Title: Polyclonal Anti-T-Lymphocyte Globulin (ATG) in Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: KD CD IKEM 1; NB/6541-3 IGA MZCR
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2004-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes mellitus; Immune intervention; Polyclonal antibodies; Type 1 diabetes of recent onset; C-peptide level 0.3 pmol/l or higher; Positivity of at least one marker of autoimmunity (diabetes)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

INTERVENTIONS:
Drug: Polyclonal anti-T-cell antibodies

SUMMARY:
The primary objective of the study is:

* To compare the effect of ATG treatment together with intensified insulin therapy (Group 1) on fasting and glucagon-stimulated C-peptide production with that of intensified insulin therapy only (Group 2) in type 1 diabetes mellitus of recent onset

Secondary objectives are:

* To compare the insulin doses between the two groups at 6, 12, 18, and 24 months after diabetes onset
* To compare the course of the specific humoral markers of autoimmunity between the groups
* To evaluate the significance of in vitro testing of specific T-cell activation by an autoantigen in the long-term follow-up in type 1 diabetes
* To assess the safety of ATG treatment in type 1 diabetes

DETAILED DESCRIPTION:
This is a randomized, controlled, single-blind and parallel group study. After admission to the hospital, initial physical and laboratory examinations will be performed. Laboratory tests and medical treatment not related to the experimental protocol (except for immunosuppressive drugs) will be performed as clinically needed. Patients who fulfill the inclusion criteria and give their informed consent to participate in the study will be randomized to be treated either with a course of ATG-Fresenius together with intensified insulin therapy (Group 1) or with intensified insulin therapy only (Group 2).

For the study purpose, clinical and laboratory status of the patients will be assessed at 14 occasions (screening, visit 1 - visit 14). Thereafter, an extended follow-up study is planned with evaluations every 6 months.

Patients will be referred to the research institution by cooperating general practitioners and diabetes specialists, preferably before initiation of insulin therapy. After diabetes confirmation (according to WHO criteria) and initial clinical and biochemical examinations (typical for all patients with recent onset diabetes) the purpose, potential risk and benefits and the design of the study will be explained. Subjects willing to participate in the study will be asked to give their written informed consent.

All patients will be actively educated in diabetes management and intensified insulin therapy (3 - 4 daily injections of human insulin, glucose self-monitoring) will be initiated according to individual needs. In subjects randomized to Group 1, 4 doses of ATG Fresenius (first dose of 9 mg/kg of body weight, then 3 consecutive doses of 3 mg/kg) will be administered intravenously over 4 hours. Subjects in Group 2 will be treated with saline infusion (500 ml) on the same days. 1 hour before the first ATG administration, a cutaneous tolerance test (0.2 ml of the final solution) will be performed. Approximately 10 days after admission the patients will be dismissed. Besides scheduled ambulant visits, all subjects will be followed-up as clinically needed. In Paediatric patients (age 15-18 years), recommendations of a paediatric endocrinologist concerning diabetes management will be respected.

After completion of the study each patient's diabetes specialist will be acquainted with the course of the treatment so far and the patients will be treated according to individual needs. They will be seen regularly once per year in the Department of Diabetes in IKEM for the next 3 years.

Discontinuation of the study:

Participation in the study may be at all times stopped according to the patient's will. Should this require the medical status of the patients, the study may be interrupted based on the investigator's decision during the period of ATG administration.

Study population:

Twenty four patients with type 1 diabetes mellitus of recent onset will be followed in the Institute for Clinical and Experimental Medicine in Prague. Inclusion criteria will be:

* Type 1 diabetes mellitus of known duration up to 6 weeks
* Men and women 15 - 35 years old, body mass index up to 32 kg/m2, exclusion of gravidity in women
* Insulin dose up to 40 IU per day for no longer than 1 month
* C-peptide level ≥ 0.3 pmol/ml 4 min. following iv. administration of 1 ml glucagon
* No previous immunosuppressive therapy, no concurrent severe infection, granulocyte count ≥ 2 x 10^9/l, platelet count ≥ 120 x 10^9/l

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Body mass index up to 32 kg/m2
* Exclusion of gravidity in women
* Known diagnosis of diabetes of less than 6 weeks
* Insulin dose of up to 40 IU per day for no longer than 1 month
* Positive for at least one autoantibody (GAD, IA2, ICA)
* C-peptide level ≥ 0.3 pmol/ml 4 min. following intravenous (IV) administration of 1 ml glucagon
* No concurrent severe infection
* Granulocyte count ≥ 2 x 10^9/l
* Platelet count ≥ 120 x 10^9/l

Exclusion Criteria:

* Other non-diabetes related autoimmune disease
* Previous immunosuppressive therapy
* Any clinical impairment precluding immunosuppressive therapy
* Leucopenia or thrombocytopenia

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28
Dates: Start 2000-11; Study Completion 2007-12

PRIMARY OUTCOMES:
C-peptide production

SECONDARY OUTCOMES:
Diabetes remission rate
Insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Frantisek Saudek, MD., Study Chair — Institute for Clinical and Experimental Medicine, Prague
Locations (1):
- Institute for Clinical and Experimental Medicine, Department of Diabetes, Prague, Czechia

REFERENCES:
- [Result] Saudek F, Havrdova T, Boucek P, Karasova L, Novota P, Skibova J. Polyclonal anti-T-cell therapy for type 1 diabetes mellitus of recent onset. Rev Diabet Stud. 2004 Summer;1(2):80-8. doi: 10.1900/RDS.2004.1.80. Epub 2004 Aug 10. PMID 17491669